CLINICAL TRIAL: NCT05742074
Title: The Effect of Faecal Microbiota Transplantation (FMT) on Eradication of Multidrug Resistant Organisms (MRO) in Intestinal Carriers - a Multicentre, Randomized, Double-blinded and Placebo-controlled Study
Brief Title: The Effect of Faecal Microbiota Transplantation (FMT) on Eradication of Multidrug Resistant Organisms (MRO) in Intestinal Carriers
Acronym: FEMRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-22040517
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Multidrug Resistant Organisms; Faecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (faecal microbiota transplantation) (Experimental): 25-30 capsules of faecal material.
  Interventions: Other: Faecal microbiota transplantation
- Placebo (Placebo Comparator): 25-30 placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Faecal microbiota transplantation — 25-30 capsules of faecal material
  Arms: FMT (faecal microbiota transplantation)
Other: Placebo — 25-30 placebo capsules
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of faecal microbiota transplantation (FMT) on eradication of multidrug resistant organisms (MRO) in the intestine. Ultimately, it would be possible to prevent invasive infections with MRO that are difficult to treat and require last-resort antibiotics. The investigators hypothesize that FMT induce intestinal resistance towards colonization with MRO e.g. Vancomycin resistant Enterococcus Faecium (VRE), carbapenemase-producing Enterobacterales (CPE) and extended-spectrum beta-lactamase producing Enterobacterales (ESBL-E).

DETAILED DESCRIPTION:
The study is designed as a randomized, double-blinded and placebo-controlled clinical trial. The participants (n = 80) will be randomized 1:1 to FMT or placebo. FMT or placebo consist of 25-30 capsules which need to be consumed on one day or alternatively consumed over three consecutive days, if one day is unacceptable to the participant. At baseline, eight weeks, and 16 weeks rectal swabs for PCR and culture will be taken. Regarding VRE and CPO, there are specific PCRs followed by confirmatory culture, whereas ESBL-E is detected by culture of rectal swab. Furthermore, participants will be asked to deliver faecal samples as well at baseline and 16 weeks post FMT to examine changes in the intestinal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Age: minimum 18 years
* Positive rectal PCR and/or culture for MRO
* Ability to speak and understand Danish or English
* Capable of swallowing the capsules

Exclusion Criteria:

* Current invasive infection with an MRO e.g. in abdomen, bloodstream or symptomatic urinary tract infection.
* Severe immune deficiency (defined as current chemo treatment or neurofilocytes < 1000/mm3
* Pancreatitis, defined by pancreatic amylases above the upper reference limit
* Planned or recent abdominal surgery (within 14 days)
* Parenteral nutrition
* Current antibiotic treatment of the same MRO as intestinal carriage
* Terminal disease with expected survival under three months
* Sepsis defined according to Surviving Sepsis Campaign guidelines
* Pregnant or lactating women

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MRO clearance | 8 weeks
  Number of participants with MRO clearance after eight weeks. This will be measured on rectal samples that will undergo PCR/culture for ESBL, VRE and CPO. The results from the test will be positive or negative.

SECONDARY OUTCOMES:
Number of participants with MRO clearance | 16 weeks
  Number of participants with negative PCR for MRO on rectal swab and faecal culture negative for MRO after 16 weeks. This will be measured on rectal samples that will undergo PCR/culture for ESBL, VRE and CPO. The result from the test will be positive or negative
Number of participants with adverse events. | 8 weeks, 16 weeks and 6 months.
  Number of participants with adverse events both severe and non-severe.
Comparison of the frequency of invasive infections | 6 months
  Comparison of the frequency of invasive infections with the same MRO as the intestinal carriage between the FMT and the placebo group.
Comparison of mortality rates, frequency of hospitalization and isolation between the FMT and the placebo group. | 6 months
  Comparison of mortality rates, frequency of hospitalization and isolation between the FMT and the placebo group.
Comparison of changes in the diversity of the intestinal microbiome between the FMT group and the placebo group. | 8 weeks and 16 weeks
  Comparison of changes in the diversity of the intestinal microbiome between the FMT group and the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Copenhagen University, Hvidovre, Copenhagen, Denmark